CLINICAL TRIAL: NCT01875939
Title: Phase-I Randomized, Open Label, Crossover Food-Effect and Absolute Bioavailability Study of WCK 2349 and WCK 771 in Healthy Adult Human Volunteers
Brief Title: Phase I, Open Label,Crossover Food-Effect and Absolute Bioavailability Study of WCK2349 and WCK771 in Healthy Adult Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: W 771/2349-101
Record Dates: First submitted 2013-05-30; First posted 2013-06-12 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Effect of Food
Keywords: healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral WCK 2349 fed/fasting (Other): This is a single center, randomized, open label, 2X2 oral IV cross over, food-effect and absolute bioavailability study. The study will be conducted in three parts i.e., Period 1 and Period 2 (foodeffect study) and Period 3 (absolute bioavailability study).
  Interventions: Drug: Oral WCK2349
- IV WCK771 (Other): This is a single center, randomized, open label, 2X2 oral IV cross over, food-effect and absolute bioavailability study. The study will be conducted in three parts i.e., Period 1 and Period 2 (foodeffect study) and Period 3 (absolute bioavailability study).
  Interventions: Drug: IV WCK771

INTERVENTIONS:
Drug: Oral WCK2349 — The subjects will be randomly assigned to receive WCK 2349 1000 mg as an oral dose in fed or fasting state (1:1) in the food effect study as per the randomization schedule. The subjects completing the food effect study (i.e., Period 1 and Period 2) will be administered WCK 771 800 mg as an intravenous infusion in fasting state in Period 3 of the study.
  Arms: Oral WCK 2349 fed/fasting
Drug: IV WCK771 — The subjects will be randomly assigned to receive WCK 2349 1000 mg as an oral dose in fed or fasting state (1:1) in the food effect study as per the randomization schedule. The subjects completing the food effect study (i.e., Period 1 and Period 2) will be administered WCK 771 800 mg as an intravenous infusion in fasting state in Period 3 of the study.
  Arms: IV WCK771

SUMMARY:
This study is aimed to ascertain the effect of food on pharmacokinetics of WCK 2349 and determine the absolute bioavailability of WCK 2349 1000 mg (oral, QD dose) with respect to WCK 771 800 mg (intravenous, QD dose).

This study would ascertain/confirm the therapeutically equivalent oral and IV doses of WCK 2349 and WCK 771 respectively, and provide guidance in case of switch over therapy (WCK 771, IV to WCK 2349, oral) in future clinical trials in patients.

DETAILED DESCRIPTION:
All the subjects will be checked-in into the clinical study facility on Day -1, the day prior to dosing. The subjects will be randomly assigned to receive WCK 2349 1000 mg as an oral dose in fed or fasting state (1:1) in the food effect study as per the randomization schedule. The subjects completing the food effect study (i.e., Period 1 and Period 2) will be administered WCK 771 800 mg as an intravenous infusion in fasting state in Period 3 of the study. There will be a washout period of three days between each period. The subjects will continue to remain in the clinical facility for the entire duration of the study (completion of three periods in the study), including wash out period. Prior to check out procedure, detailed clinical examination will be done to confirm that subject has no safety issues.

ELIGIBILITY:
Inclusion Criteria:

* If female, postmenopausal for at least 1 year,surgically sterile or birth control measures.
* Body Mass Index (BMI) between 18 and 32
* No significant diseases
* No recent history of smoking or alcohol

Exclusion Criteria:

* Known history of hypersensitivity or idiosyncratic reaction to quinolones or any other related drugs.
* History or evidence of disease or condition which might compromise the haemopoietic, renal, hepatic,endocrine, pulmonary, central nervous, cardiovascular,immunological, dermatological, gastrointestinal or any other body system.
* No receipt of a prescription drug or non-prescription drug .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate pharmacokinetics of WCK 2349 (Fed/Fasting)and WCK 771 Fasting | Approximately 11 days
  To compare the pharmacokinetics of WCK 2349 following oral administration of 1000 mg of WCK 2349 (QD, one day) in healthy, adult, human subjects in fed and fasting state To determine the absolute bioavailability of WCK 2349 following oral administration of 1000 mg of WCK 2349 (QD, one day) with respect to intravenous administration of 800 mg of WCK 771 (QD, one day) in healthy adult human subjects in fasting state.Absolute bioavailability (F) of oral WCK 2349 as compared to intravenous WCK 771 following single dose administration in healthy subjects in fasting state will be calculated as follows: F =AUC i.v /AUC oral *Dose of oral/Dose of IV Summary statistics will be provided for the safety data.

SECONDARY OUTCOMES:
safety of oral WCK 2349 and intravenous WCK 771 in healthy adult human subjects | Approximately 11 days
  Safety assessed by physical, clinical examination, vital sign, laboratory test, ECG recordings and adverse event recording at EOT visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha A Mondal, MD, Principal Investigator — PPD Phase I unit
Locations (1):
- PPD Phase I unit, 7551 Metro Center Drive, Suite 200, Austin, Texas, United States